CLINICAL TRIAL: NCT03750058
Title: AXONE -Acute : Acute Assessment of a Micro Multipolar Lead for Enhanced Cardiac Resynchronisation Therapy
Brief Title: Acute Assessment of a Micro Multipolar Lead for Enhanced Cardiac Resynchronisation Therapy
Acronym: AXONE-Acute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017/170/HP
Record Dates: First submitted 2018-07-27; First posted 2018-11-21 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Resynchronisation Therapy
Keywords: quadripolar LV leads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant test procedure (Experimental): Implant test procedure with new LV quadripolar lead before a standard implantation for Cardiac resynchronisation therapy
  Interventions: Device: Implant test procedure

INTERVENTIONS:
Device: Implant test procedure — Implant test procedure with new LV quadripolar lead before a standard implantation for Cardiac resynchronisation therapy

SUMMARY:
Pilot study to evaluate the performance of a lead below 2 French with specific distal shape to deliver efficient LV pacing

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥18 years old.
* Patient presenting a CRT-P or CRT-D indication according to the latest ESC guidelines .
* Primary implant of a CRT device (including upgrade from a single or dual-chamber pacemaker or ICD).
* Signed and dated informed consent.
* Patient affiliated with, or beneficiary of a social security category.

Exclusion Criteria:

* Class IV of NYHA (ambulatory or not).
* Allergy to contrast media used for imaging during cardiac catheterization.
* Severe Renal Failure (clearance of creatinine < 30ml/mn/m²).
* Previous failure catheterization of the coronary sinus, or previous failure of left ventricular lead implantation.
* Already included in another clinical study involving intra-cardiac active implantable device, or participation to any other clinical trial in the last 2 weeks.
* Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision).
* Known pregnancy, breastfeeding women or in childbearing age without an adequate contraceptive method (failure rate < 1%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
LV Multizone pacing success rate | 20 min
  Percent of patients where the placement of the AXONE lead provides two distant LV pacing vectors matching Pacing Threshold ≤ 3.5V/0.5ms
LV pacing success rate | 20 min
  Percent of patients where the placement of the AXONE lead allows at least one LV pacing vector matching Pacing Threshold ≤ 3.5V/0.5ms

SECONDARY OUTCOMES:
Implant testing Procedure-related Adverse Events procedure. | 1 month post testing
Electrical performance of device (1) | 20 min
  Electrical performance focusing on LV pacing threshold (Volts)
Electrical performance of device (2) | 20 min
  Electrical performance focusing on LV pacing impedance (Ohm)
Lead Implant Efficiency | 20 min
  procedure time for successful placement
Lead Implant Efficiency | 20 min
  Radiation dose during implant
Satisfaction of implanter | 20 min
  handling assessment of implanter using satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ANSELME, Pr, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - Bordeaux University Hospital, Bordeaux
  - Lille University Hospital, Lille
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No